CLINICAL TRIAL: NCT04412863
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of VIR-2218 Alone or in Combination With Pegylated Interferon Alpha-2a
Brief Title: Study of VIR-2218 With or Without Pegylated Interferon Alpha-2a for Treatment of Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-2218-1001-PEG-IFNα
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Cohort 1d (Experimental): VIR-2218 given by subcutaneous injection
  Interventions: Drug: VIR-2218
- Cohort 2d (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 3d (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 1e (Experimental): VIR-2218 given by subcutaneous injection
  Interventions: Drug: VIR-2218
- Cohort 2e (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 3e (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 1f (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 2f (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a
- Cohort 3f (Experimental): VIR-2218 and pegylated interferon-alfa 2a given by subcutaneous injection
  Interventions: Drug: VIR-2218; Drug: pegylated interferon-alfa 2a

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection
Drug: pegylated interferon-alfa 2a — pegylated interferon-alfa 2a given by subcutaneous injection
  Other Names: pegylated interferon alpha-2a; PEG-IFNα
  Arms: Cohort 1f; Cohort 2d; Cohort 2e; Cohort 2f; Cohort 3d; Cohort 3e; Cohort 3f

SUMMARY:
This is a phase 2 study in which subjects with chronic hepatitis B virus (HBV) infection will receive VIR-2218 alone or in combination with pegylated interferon alfa-2a and will be assessed for safety, tolerability, pharmacokinetics, and antiviral activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of ages 18 - 65
* Chronic HBV infection for >/= 6 months

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* Significant fibrosis or cirrhosis
* History or evidence of drug or alcohol abuse
* History of intolerance to SC injection
* History of chronic liver disease from any cause other than chronic HBV infection
* History of hepatic decompensation
* Any prior receipt of an interferon product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events as assessed by CTCAE v5.0 | Up to 148 Weeks
Number of subjects with abnormalities in vital signs, electrocardiogram (ECG), and clinically significant laboratory findings | Up to 148 Weeks

SECONDARY OUTCOMES:
Mean maximum reduction of serum HBsAg at any timepoint | Up to 144 Weeks
Number of subjects with serum HBsAg loss (undetectable HBsAg) at any timepoint | Up to 144 Weeks
Number of subjects with sustained serum HBsAg loss (undetectable HBsAg) for greater than 6 months | Up to 144 Weeks
Number of subjects with anti-HBs seroconversion at any timepoint | Up to 144 Weeks
For HBeAg-positive subjects: number of subjects with HBeAg loss (undetectable HBeAg) and/or anti-HBe seroconversion at any timepoint | Up to 96 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Australia (2):
  - Investigative Site, Birtinya, Queensland
  - Investigative Site, Fitzroy, Victoria
- Investigative site, Hong Kong, Hong Kong
- Malaysia (4):
  - Investigative Site, Batu Caves
  - Investigative Site, Kajang
  - Investigative Site, Kuala Lumpur
  - Investigative Site, Kuantan
- Investigative Site, Auckland, New Zealand
- South Korea (5):
  - Investigative Site, Busan
  - Investigative Site, Chuncheon
  - Investigative Site, Daegu
  - Investigative Site, Seoul
  - Investigative Site, Yangsan
- Thailand (5):
  - Investigative Site, Bangkok
  - Investigative Site, Chiang Mai
  - Investigative Site, Hat Yai
  - Investigative Site, Khlong Luang
  - Investigative Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: No